CLINICAL TRIAL: NCT03977272
Title: Comparison of Therapeutic Effect Between Combination of Anti-PD-1 Antibody With mFOLFIRINOX and mFOLFIRINOX Alone in Metastatic Pancreatic Cancer Patients: A Randomized Clinical Trial
Brief Title: Combination of Anti-PD-1 Antibody and Chemotherapy in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Proffessor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CISPD3
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Anti-PD-1 Antibody
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Combinations; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy group (Active Comparator): Treatment with modified-FOLFIRINOX Folic acid 400mg/m^2, 5- fluorouracil 2400mg/m^2 for 46h, irinotecan 135mg/m^2 and oxaliplatin 68mg/m^2
  Interventions: Drug: Chemotherapy
- Combination group (Experimental): Treatment with modified-FOLFIRINOX and Anti-PD-1 antibody Folic acid 400mg/m^2, 5- fluorouracil 2400mg/m^2 for 46h, irinotecan 135mg/m^2 and oxaliplatin 68mg/m^2, Anti-PD-1 antibody 200mg.
  Interventions: Drug: Combination drug

INTERVENTIONS:
Drug: Combination drug — Accompanying with modified-FOLFIRINOX, Anti-PD-1 antibody was applied biweekly
  Arms: Combination group
Drug: Chemotherapy — modified-FOLFIRINOX
  Arms: Chemotherapy group

SUMMARY:
The prognosis of pancreatic cancer is extremely poor. NCCN guidelines recommend FOLFIRINOX or modified-FOLFIRINOX as the first-line chemotherapeutic regimen. Studies have shown that immunotherapy with Anti-PD-1 antibody can effectively increase the response rate and prolong patient survival in a number of cancer diseases. Here investigators intend to compare the therapeutic effects of modified-FOLFIRINOX alone and the combination of modified-FOLFIRINOX and Anti-PD-1 antibody in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Metastatic pancreatic cancer patients will be enrolled in this trial. Investigators will assign patients to the treatment after randomization. The primary endpoint is overall survival. Response rate, progression-free survival, drugs related side effects and other endpoints events will be recorded and analyzed, to assess the combination treatment with modified-FOLFIRINOX and Anti-PD-1 antibody could or couldn't benefit the patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* •Pathologically (histologically or cytologically) confirmed pancreatic ductal adenocarcinoma (PDAC).

  * Recurrent disease or metastatic disease (such as liver, peritoneum, lung) evaluated by abdominal contrast-enhanced CT, MRI, and chest CT. PET/CT or other imaging examinations would be used if necessary.
  * Never receive any systematic treatment or Progression after fisrt line Gemcitabine base chemotherapy
  * ECOG score 0 or 1.
  * Serum creatinine level is normal, and serum total bilirubin level is less than 1.5 x ULN.
  * ALT and AST are less than 2 x ULN.
  * Signed informed consent.

Exclusion Criteria:

* •History of participation of other clinical trails within 4 weeks

  * History of autoimmune disease or other condition receiving glucocorticoid treatment
  * History of receiving chemotherapy within 2 weeks
  * History of radiotherapy and molecular target therapy within 2 weeks
  * History if active tuberculosis
  * History of malignance treatment in the past, excluding basal and cutaneous squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma
  * Major cardiovascular diseases (including myocardial infarction, unstable angina, congestive heart failure, severe uncontrolled arrhythmia) during the past six months of enrollment.
  * Hematological precancerous diseases, such as myelodysplastic syndromes.
  * Evidence of clinical-related or previous interstitial lung disease, such as noninfectious pneumonia or pulmonary fibrosis, or baseline chest CT scan or chest X-ray findings
  * Previous or physical findings of central nervous system disease, except for adequately treated (e.g. primary brain tumors, uncontrolled seizures or strokes with standard medications)
  * Preexisting neuropathy > 1 (NCI CTCAE).
  * Immune deficiency syndrome, such as active tuberculosis and HIV infection.
  * Allograft requires immunosuppressive therapy or other major immunosuppressive therapies.
  * Severe serious wounds, ulcers or fractures.
  * Clinical evaluation is unacceptable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Through the study peirod, for 3 years
  The period from the first study treatment to any cause of death

SECONDARY OUTCOMES:
Resection rate | Through the study peirod, for 3 years
  The number of cases received surgery / the total number of evaluable cases (%)
Objective response rate | Through the study peirod, for 3 years
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%)
Disease control rate | Through the study peirod, for 3 years
  The number of cases in which response (PR + CR) and stable disease (SD) are achieved from the start of cell infusion/the total number of evaluable cases (%)
Progression-free survival | Through the study peirod, for 3 years
  The period from the first treatment to the first evaluation of PD or any cause of death
Adverse effects | Through the study peirod, for 3 years
  Adverse events occurring through the study treatment, such as abnormalities or changes in laboratory examinations, physical examinations, vital signs, etc.
Carbohydrate antigen 19-9 | Through the study peirod, for 3 years
  The change of CA 199
EORTC QLQ - PAN26 score | Through the study peirod, for 3 years
  The change of the quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fu Q, Chen Y, Huang D, Guo C, Zhang X, Xiao W, Xue X, Zhang Q, Li X, Gao S, Que R, Shen Y, Wu J, Zhang M, Bai X, Liang T. Sintilimab Plus Modified FOLFIRINOX in Metastatic or Recurrent Pancreatic Cancer: The Randomized Phase II CISPD3 Trial. Ann Surg Oncol. 2023 Aug;30(8):5071-5080. doi: 10.1245/s10434-023-13383-w. Epub 2023 Apr 13. PMID 37052821